CLINICAL TRIAL: NCT05848765
Title: Relapsed Follicular Lymphoma Randomised Trial Against Standard ChemoTherapy (REFRACT): A Randomised Phase II Trial of Investigator Choice Standard Therapy Versus Sequential Novel Therapy Experimental Arms
Brief Title: Relapsed Follicular Lymphoma Randomised Trial Against Standard ChemoTherapy
Acronym: REFRACT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Cancer Research UK (Other); Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RG_22-020
Record Dates: First submitted 2023-04-18; First posted 2023-05-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Relapsed Follicular Lymphoma; Refractory Follicular Lymphoma
Keywords: Epcoritamab; Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — Lenalidomide; Rituximab; obinutuzumab; Bendamustine Hydrochloride; Vincristine; Doxorubicin; Cyclophosphamide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Round 1: Epcoritamab and lenalidomide (Experimental): Epcoritamab (weekly for cycles 1 and 2 and on day 1 of cycles 3-12 for up to 12 cycles) and lenalidomide (daily for days 1-21 of each cycle for up for 12 cycles), cycles will be 28 day cycles.
  Interventions: Drug: Epcoritamab; Drug: Lenalidomide
- Round 2 (Experimental): Investigation agent 2
  Interventions: Drug: Investigation agent 2
- Round 3 (Experimental): Investigation agent 3
  Interventions: Drug: Investigation agent 3
- All rounds: Investigator Choice Therapy (Active Comparator): Choice of therapy to be selected by the Investigator for each patient prior to randomisation. The Investigator will choose between; RCHOP, RCVP, rituximab and bendamustine, rituximab and lenalidomide or bendamustine and obinutuzumab.
  Interventions: Drug: Lenalidomide; Drug: Rituximab; Drug: Obinutuzumab; Drug: Bendamustine; Drug: Vincristine; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Prednisone

INTERVENTIONS:
Drug: Epcoritamab — Bispecific antibody
  Arms: Round 1: Epcoritamab and lenalidomide
Drug: Lenalidomide — Immunomodulatory agent
  Arms: All rounds: Investigator Choice Therapy; Round 1: Epcoritamab and lenalidomide
Drug: Rituximab — Monoclonal antibody
  Arms: All rounds: Investigator Choice Therapy
Drug: Obinutuzumab — Monoclonal antibody
  Arms: All rounds: Investigator Choice Therapy
Drug: Bendamustine — Alkylating agent (chemotherapy drug)
  Arms: All rounds: Investigator Choice Therapy
Drug: Vincristine — Antineoplastic, Vinca Alkaloid
  Arms: All rounds: Investigator Choice Therapy
Drug: Doxorubicin — Anthracycline
  Arms: All rounds: Investigator Choice Therapy
Drug: Cyclophosphamide — Alkylating agent (chemotherapy drug)
  Arms: All rounds: Investigator Choice Therapy
Drug: Prednisone — Corticosteroid
  Arms: All rounds: Investigator Choice Therapy
Drug: Investigation agent 2 — The drug used in round 2 is yet to be confirmed, round 2 is estimated to open in Q4 2025 and the record will be updated when the drug has been confirmed
  Arms: Round 2
Drug: Investigation agent 3 — The drug used in round 3 is yet to be confirmed, round 3 is estimated to open in Q3 2027 and the record will be updated when the drug has been confirmed
  Arms: Round 3

SUMMARY:
The aim of the REFRACT clinical trial is to find new therapies with improved outcomes compared to the current standard treatment available, in patients with relapsed or refractory follicular lymphoma. This will be done by comparing patients who have received a new treatment against patients who receive standard treatment based on their response to the treatment received.

DETAILED DESCRIPTION:
In the REFRACT trial patients with relapsed or refractory follicular lymphoma (rrFL) will be randomised (randomly allocated) to receive a new treatment (experimental treatment) or standard treatment which will be chosen by their doctor prior to entering the trial (called investigator choice standard therapy (ICT)). There are 3 treatment rounds which will happen one after another, testing 3 different experimental treatments. The experimental treatment in each round will be compared to ICT. ICT will be a choice of 1 of 5 standard treatment options including RCHOP, RCVP, lenalidomide and rituximab, bendamustine and rituximab or obinutuzumab and bendamustine. Patients in Round 1 (R1) will be randomised using a 1:1 allocation ratio (meaning patients have a 50/50 chance of receiving the experimental treatment). In Round 1 the experimental treatment is epcoritamab combined with lenalidomide. Patients randomised to epcoritamab and lenalidomide will receive up to 12 28-day cycles of therapy; epcoritamab will be delivered as a subcutaneous injection weekly for cycles 1 and 2 and on day 1 of cycles 3-12. Lenalidomide will be taken orally on days 1-21 of each cycle. Patients in Rounds 2 (R2) and 3 (R3) (experimental treatments yet to be determined) will be randomised using a 1:4 allocation ratio in favour of the experimental treatment (meaning patients are more likely to receive the experimental treatment). The study will recruit 284 patients with rrFL over 5 years. The aim is to identify new therapies which have better outcomes compared to ICT based on patients response to treatment (tested by PET scan) after 24 weeks of therapy. Following treatment patients will be followed up yearly until the end of the trial (up to 10 years).

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven relapsed or refractory CD20 positive, grade 1-3a follicular lymphoma (biopsy within 3 months of trial entry)
2. Aged 18 years or over
3. Advanced disease that in the opinion of the treating physician requires treatment
4. Patient suitable for standard available therapy at the Investigator's discretion
5. Prior therapy with at least one line of immunochemotherapy. Previous radiotherapy at any time is permitted and will not count as a line of therapy. Previous rituximab monotherapy is also permitted as long as patients have at any time also received at least one line of immunochemotherapy
6. Assessable disease by PET-CT (at least one involved node with long diameter >1.5cm, or extranodal lesion >1cm )
7. ECOG performance status of 0, 1 or 2 at trial entry
8. Adequate organ function defined as; i. ANC ≥ 1.0 x 109/L (growth factor use is permitted) ii. Platelet count ≥ 75 x 109/L, or ≥ 50 x 109/L if bone marrow infiltration or splenomegaly iii. ALT and AST level ≤3 x ULN iv. Direct bilirubin level ≤ 2 x ULN, unless due to Gilbert's syndrome v. CrCl ≥ 50mL/min (by Cockcroft-Gault formula) vi. PT, INR and aPTT ≤ 1.5 x ULN, unless receiving anticoagulation vii. LVEF within normal limits by MUGA or echocardiography
9. Able to provide written informed consent
10. Women of childbearing potential (or their partners) must use an effective form of contraception

Exclusion Criteria:

1. Current (or within 1 year) transformation to high grade lymphoma, including grade 3b follicular lymphoma (patients with historical high-grade transformation over 1 year ago are eligible)
2. Non-Fluorodeoxyglucose (FDG) avid disease
3. Prior allogenic stem cell transplantation (SCT) or solid organ transplant
4. Prior treatment with lenalidomide
5. Treatment with CAR-T therapy within 100 days of starting trial treatment
6. SCT or maintenance therapy planned within 24 weeks of starting treatment (patients planning SCT/maintenance after at least 24 weeks of treatment are eligible)
7. Immunochemotherapy with a platinum-containing regimen planned
8. Known serological positivity for HIV or uncontrolled HCV
9. Hepatitis B surface antigen (HBsAg) positive and/or detectable viral DNA. Patients positive for Hepatitis B core antibody (anti-HBc) but viral DNA negative are eligible
10. Other malignancy within 2 years of enrolment, excepting cervical carcinoma stage 1B or less, non-invasive basal cell or squamous cell skin carcinoma, non-invasive, superficial bladder cancer, prostate cancer with a current PSA level <0.1ng/mL, any curable cancer with a CR of > 2 years duration
11. Active systemic infection requiring treatment
12. Current or prior CNS involvement with lymphoma
13. History of allergy or anaphylaxis to anti-CD20 monoclonal antibody therapy
14. Known hypersensitivity to any of the experimental arm IMPs. Patients with a known hypersensitivity to a control arm regimen may still be eligible if they have no hypersensitivity to other potential control arm IMPs.
15. Serious medical or psychiatric illness likely to interfere with participation in this clinical study
16. Recent cancer treatment (chemotherapy, immunotherapy, biological therapy) within 4 weeks of starting trial treatment; systemic steroid treatment (prednisolone > 10mg daily (or equivalent)) within 7 days of cycle 1 day 1 dosing
17. Unwilling to use appropriate contraception methods whilst on study treatment and for 12 months following end of treatment (or 18 months for female patients whose ICT regimen contains obinutuzumab)
18. Women who are pregnant or breastfeeding
19. Prior treatment with the experimental therapy under investigation
20. Major surgery within 30 days of starting treatment
21. Severe arrhythmias, heart failure, previous myocardial infarction, acute inflammatory heart disease for ICT regimen containing doxorubicin, or severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease for ICT regimen containing rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Complete metabolic response (CMR) | 24 weeks
  CMR will be assessed by PET-CT using the Deauville 5-point scale and Lugano 2014 criteria. Patients who die from any cause or relapse/progress prior to this time-point will be considered non-responders. Patients who don't have a PET-CT scan within the protocol defined window or withdraw from the trial prior to this time-point will be considered non outcome evaluable. Patients who undergo stem-cell transplant (SCT) within 24 weeks of randomisation, patients who fail to start treatment and patients whose ineligibility is deemed to impact upon response to treatment will be replaced and hence not included in the analysis of this outcome

SECONDARY OUTCOMES:
Overall metabolic response | 24 weeks
  Complete metabolic response (CMR) and partial metabolic response (PMR) will be assessed by PET-CT. Patients who die from any cause or relapse/progress prior to this time-point will be considered non-responders. Patients who undergo stem-cell transplant (SCT) within 24 weeks of randomisation, patients who fail to start treatment and patients whose ineligibility is deemed to impact upon response to treatment will be replaced and hence not included in the analysis of this outcome
Progression free survival (PFS) | 10 years
  The time from randomisation to the date of first disease progression or death. Patients who are alive and relapse/progression at the time of analysis will be censored at their date last seen
Overall survival (OS) | 10 years
  The time from randomisation to the date of death from any cause. Patients who are alive at the time of analysis will be censored at their date last seen
Duration of response (DoR) | 10 years
  The time from complete and partial metabolic response by PET-CT to relapse/progression or death from any cause. Patients who are alive and relapse/progression free at the time of analysis will be censored at their date last seen
Duration of complete response (DoCR) | 10 years
  The time from complete metabolic response by PET-CT to relapse/progression or death from any cause. Patients who are alive and relapse/progression free at the time of analysis will be censored at their date last seen
Time to next treatment (TTNT) | 10 years
  The time from randomisation to the start date of next treatment for lymphoma. Patients who are responding (CMR or PMR) who receive consolidation radiotherapy will not be considered an event and will be censored at their date last seen if no other treatment for lymphoma is reported. Patients who die without having started next lymphoma treatment will be considered a competing risk at their date of death, and patients who are alive and have not started next lymphoma treatment at the time of analysis will be censored at their date last seen
Adverse events (AEs) | Collected from start of treatment until 60 days after treatment
  Collected and reported in accordance with CTCAE version 5 defined as the number of patients who experience one or more grade 3 or 4 adverse events or serious adverse events of any grade
Quality of Life (QoL) | Collected pre-treatment, day 1 of cycle 3 (28 day cycles), 24 weeks from treatment start and then every 24 weeks in non-progressed patients until the end of the study (10 years)
  Measured using the EQ-5D-5L and FACT-Lym
Quality of Life (QoL) | Collected pre-treatment, day 1 of cycle 3 (28 day cycles), 24 weeks from treatment start and then every 24 weeks in non-progressed patients until the end of the study (10 years)
  Measured using the FACT-Lym

CONTACTS AND LOCATIONS:
Locations (25):
- United Kingdom (25):
  - NHS Grampian, Aberdeen
  - Belfast Health & Social Care Trust, Belfast
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and vale University LHB, Cardiff
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Croydon Health Services NHS Trust, Croydon
  - NHS Greater Glasgow and Clyde, Glasgow
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - University Hospital of North Midlands NHS Trust, Stoke-on-Trent
  - Swansea Bay University Local Health Board, Swansea
  - Torbay and South Devon NHS Foundation Trust, Torquay

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaskell C, Linton K, Bishton M, McIlroy G, Lax S, Fox S, Hopkins L, Collings R, Rhodes M, Seale T, Jackson A. The REFRACT trial: implementation of Bayesian power priors in a randomised, sequential phase II adaptive platform trial. BMC Med Res Methodol. 2025 May 3;25(1):121. doi: 10.1186/s12874-025-02575-5. PMID 40319227
- [Derived] McIlroy G, Lax S, Gaskell C, Jackson A, Rhodes M, Seale T, Fox S, Hopkins L, Okosun J, Barrington SF, Ringshausen I, Ramsay AG, Calaminici M, Linton K, Bishton M. Investigator choice of standard therapy versus sequential novel therapy arms in the treatment of relapsed follicular lymphoma (REFRACT): study protocol for a multi-centre, open-label, randomised, phase II platform trial. BMC Cancer. 2024 Mar 25;24(1):370. doi: 10.1186/s12885-024-12112-0. PMID 38528445